CLINICAL TRIAL: NCT04059965
Title: AntiCoagulation Tracking InterVention and Evaluation: Using a Customized Panel Management Platform to Improve Outcomes for Patients on Anticoagulation
Brief Title: AntiCoagulation Tracking InterVention and Evaluation
Acronym: ACTIVE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P0534218
Record Dates: First submitted 2019-05-27; First posted 2019-08-16 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Anticoagulation; Atrial Fibrillation; Atrial Flutter; Pulmonary Embolus/Emboli; Deep Vein Thrombosis; Stroke; Hypercoagulability
MeSH Terms: conditions — Atrial Fibrillation; Atrial Flutter; Pulmonary Embolism; Embolism; Venous Thrombosis; Stroke; Thrombophilia

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): This cohort of patients will receive panel management through a customize software that integrates with the electronic health record
  Interventions: Other: Panel Management for Anticoagulation Therapy
- Control Arm (Active Comparator): This cohort of patients will receive usual care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Panel Management for Anticoagulation Therapy — Patients in the intervention arm will receive notifications reminding them of upcoming labs and appointments. We hypothesize this will improve adherence and therapeutic control and reduce risk for bleeds and/or strokes
  Arms: Intervention Arm
Other: Usual Care — Patients will receive standard, protocolized care in their respective anticoagulation clinics
  Arms: Control Arm

SUMMARY:
Anticoagulants are a leading cause of acute injury from adverse drug events, leading to ~20,000 serious injuries reported to the Food and Drug Administration per year and more than 220,000 emergency department visits annually. Therefore, we propose to implement a health information technology (HIT) population management tool at two distinct anticoagulation clinics that will allow the care team to assign and track tasks essential for timely patient monitoring. We will examine its effect on anticoagulation management outcomes through a randomized trial, hypothesizing that such interventions can be effective as well as cost-effective strategies to improve patient safety in the context of anticoagulation management services.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥18 years)
* those prescribed an anticoagulation medication at Zuckerberg San Francisco General Hospital or University of California, San Francisco Health

Exclusion Criteria:

* Minors (age<18)
* those not prescribed anticoagulation medication at ZSFG or UCSF Health

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Time in Therapeutic Range | 6 months
  Using the Rosendaal method, we will assess the proportion of the treatment duration that the patient's International Normalized Ratio is within the goal therapeutic range.

SECONDARY OUTCOMES:
Proportion Time in Range | 6 months
  Simple ratio of proportion of time patient's International Normalized Ratio is in goal range.
Time from initiation to therapeutic INR (TWTR) | Study Period (average of 2 years)
  Time to achieve first therapeutic international normalized ratio
Adverse events | Study Period (average of 2 years)
  Incidence of bleeds, deep vein thrombosis, pulmonary embolism, and stroke)

OTHER OUTCOMES:
Time from out-of-range to patient contact (T2C) | Study Period (average of 2 years)
  Time it takes clinicians to respond to abnormal test results
Adherence to monitoring guidelines | Study Period (average of 2 years)
  Proportion of patients who receive follow-up in a timely manner as defined by treatment guidelines
Attendance/ no-show rate | Study Period (average of 2 years)
  Rate of missed appointments
Timely discontinuation of treatment | Study Period (average of 2 years)
  Timeliness of treatment duration assessed as percentage of time on therapy in excess of what was prescribed

CONTACTS AND LOCATIONS:
Overall Officials: Urmimala Sarkar, MD, MPH, Principal Investigator — University of California, San Francisco

IPD SHARING:
Plan to Share IPD: No